CLINICAL TRIAL: NCT06835868
Title: Nationwide Dynamic Register for Screening, Evaluation and Follow-up of Patients Suffering From Chronic Pain Syndromes and Treated by Means of Invasive Neuromodulation.
Brief Title: Neuro-Pain Provides a Dynamic and Interactive Register for the Invasvive Neuromodulatory Therapies for Different Chronic Pain Syndromes. Patients Living in Belgium and Suffering From Persistent Spinal Pain Syndromes Type 2 as Well as Suffering From Complex Regional Pain Syndromes Are Included.
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: Neuro-Pain
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain Syndromes; CRPS
Keywords: spinal cord stimulation; chronic pain; quality of life
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Spinal cord stimulation — implantation of electrode which is linked to an implantable impulse generator for the treatment of chronic pain syndromes.

SUMMARY:
Patients suffereing from chronic pain due to persistent spinal pain syndromes or complex regional pain syndromes and living in Belgium will be included in this register once they are being considered for a treatment with invasive neuromodulation (either spinal cord stimulation either dorsal root ganglion stimulation). The screening process, the multidisciplinary evaluation, the trial therapy and the long-terl follow-up will be monitored through this register.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain syndromes

Exclusion Criteria:

* acute pain syndromes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients suffering from chronic pain syndromes, either persistent spinal pain syndromes or complex regional pain syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity after 21 days | 21 days
  Follow-up of pain intensity (measured by the Numeric Rating Scale, with a minimum of 0 and a maximum score of 10) during the trial therapy of 21 days, together with quality of sleep and quality of ambulation (also ona NRS scale from 0 to 10).

CONTACTS AND LOCATIONS:
Locations (1):
- UZA, multidisciplinary pain center, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bernaerts L, Roelant E, Moens M, Ly HG, Buyten JV, Billet B, Bryon B, Puylaert M, Tuna T, Malone M, Theys T, Berquin A, Vangeneugden J, Hans G. Multidisciplinary Approach to Spinal Cord Stimulation for Persistent Spinal Pain Syndromes: A 65-Month Integrated Data Collection From the Belgian Neuro-Pain(R) Real-World Data Register. Pain Res Manag. 2025 Aug 4;2025:7880611. doi: 10.1155/prm/7880611. eCollection 2025. PMID 40791635